CLINICAL TRIAL: NCT01632215
Title: Effect of Preoperative Gabapentine for Carpal Tunnel Syndrome
Brief Title: Preoperative Gabapentine for Carpal Tunnel
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Rioko Kimiko Sakata, Pain Clinic Director, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEP 0223/09
Record Dates: First submitted 2012-06-28; First posted 2012-07-02 (Estimated); Results first posted 2014-06-04 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Carpal Tunnel Syndrome
Keywords: gabapentine; postoperative pain
MeSH Terms: conditions — Carpal Tunnel Syndrome; Pain, Postoperative | interventions — Gabapentin; Anticonvulsants; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- preoperative gabapentine, (Experimental): Gabapentine
  Interventions: Drug: Gabapentine
- sugar pill (Placebo Comparator): Placebo group
  Interventions: Other: Sugar pill

INTERVENTIONS:
Drug: Gabapentine — Gabapentine 600 mg 01 dose
  Other Names: Anticonvulsant
  Arms: preoperative gabapentine,
Other: Sugar pill — Sugar pill 01 dose
  Arms: sugar pill

SUMMARY:
The purpose of this study was to evaluate the postoperative analgesic effect of preoperative gabapentine for carpal tunnel syndrome surgery.

DETAILED DESCRIPTION:
There was studied 40 patients. Group 1 patients received 600 mg of gabapentin 1 hour before surgery; G2 received placebo 1 hour before surgery.

Anesthesia was regional intravenous block. Postoperative analgesia when needed was with acetaminophen. If needed was administered codeine. The evaluation of neuropathic pain was made by DN4 questionnaire. Pain intensity was assessed by numeric scale at block and after 30min, 1h, 2h, 2wk, 4wk, 6m. It was noted the duration of analgesia, and the amount of acetaminophen and codeine.

The statistical program used for analysis of the results was the Instat Graph

ELIGIBILITY:
Inclusion Criteria:

* carpal tunnel syndrome

Exclusion Criteria:

* disorientation, psychiatric disease, myocardial ischemia, hypertension, arrhythmia, another pain syndrome, drug user, and pregnant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2011-08 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rioko K Sakata, PhD, Study Director — Universidade Federal de São Paulo

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Preoperative Gabapentine, | Sugar Pill
Started | 20 | 20
Completed | 18 | 19
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Preoperative Gabapentine, | Sugar Pill | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Median (Full Range); unit: years] — gabapentine 51,5 (41 - 59) Sugar pill 52,1 (35 - 70)
  years | 51.5 [41 to 59] | 52.1 [35 to 70] | 51.8 [35 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity
Description: Numerical score from 0 to 10; zero means no pain and 10 is the more intense pain
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Preoperative Gabapentine, | Sugar Pill
Number analyzed (Participants) | 18 | 19
units on a scale | 0.3 (0.8) | 0.4 (1.8)

2. Secondary Outcome: Chronic Pain
Description: Numerical score from 0 to 10 scale:
  Minimum value= zero (means no pain) and Maximum value= 10 (more intense pain)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Preoperative Gabapentine, | Sugar Pill
Number analyzed (Participants) | 20 | 20
points
  30 minutes after surgery | 5.5 (2.7) | 6.9 (2.5)
  1 hour after surgery | 2.4 (1.6) | 3.4 (2.9)
  2h after | 0.3 (0.8) | 0.6 (1.0)
  2 weeks after | 3.6 (3.4) | 4.6 (3.1)
  1 month after | 3.2 (3.3) | 3.6 (3.4)
  3 months after | 1.8 (3.0) | 1.6 (2.7)
  6 months after | 1.3 (2.9) | 1.2 (2.2)
Statistical Analysis 1: Comparison: Preoperative Gabapentine,; Test type: Superiority; p < 0.05, t-test, 1 sided; Mean Difference (Net) = 0.3

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Preoperative Gabapentine, | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No